CLINICAL TRIAL: NCT00300833
Title: Treating Acute MI Patients With Aggrastat on Their Way to Hospital
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Menachem Nahir, The baruch Padeh Medical center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Aggrastat in AMI.CTIL
Record Dates: First submitted 2006-03-01; First posted 2006-03-10 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2009-01

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Tirofiban

INTERVENTIONS:
Drug: Tirofiban — pci

SUMMARY:
Treating an AMI patient with ST elevation with Aggrastat in the ambulance on his or her way to the hospital.

ELIGIBILITY:
Inclusion Criteria:

patients with acute Myocardial infarction with ST elevation , and moving by ambulance to Poriya hospital

Exclusion Criteria:

* women less than 50 years old and 80 years old, bleeding tendency, stroke in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-01; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
mortality | immidiately

SECONDARY OUTCOMES:
TIMI flow | 24 hours
  feeling better

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Naheer, Study Chair — The Baruch Padeh Medicel Center, Poriya, Tiberias, Israel
Locations (2):
- Israel (2):
  - Cardiovascular Division, The Baruch Padeh Medical Center, Poriya,, Tiberias
  - Magen David ,, Tiberias